CLINICAL TRIAL: NCT02628431
Title: The Application of the ELFI-TECH Monitor for Measurement of Blood Pressure, Cardiac Output and Extend of Regional and Neuraxial Anesthesia: The Elfitor Study
Brief Title: The Application of the ELFI-TECH Monitor for Perioperative Hemodynamic Measurements
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Albert Dahan, MD, PhD, Professor, Leiden University Medical Center
Other Study IDs: P14.173
Record Dates: First submitted 2015-12-06; First posted 2015-12-11 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Colon Carcinima

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- General anesthesia: Patients that will recieve general anesthesia for elective surgery
  Interventions: Device: Elfi tech monitor
- Regional or neuraxial anesthesia: Patients that will revieve regional or neuraxial anesthesia for elective surgery
  Interventions: Device: Elfi tech monitor

INTERVENTIONS:
Device: Elfi tech monitor
  Other Names: Elfitor

SUMMARY:
The elfitor device is a small non invasive device that uses dynamic light scattering to measure skin bloodflow, blood velocity, coagulation and hemodynamic parameters. In this study, the investigators will investigate whether the elfitor device is able to detect changes in bloodpressure, cardiac output during general anesthesia. Furthermore, the investigators will investigate changes in cutanuous blood flow in different parts of the body during peripheral nerve or neuraxial block.Being able to monitor these entities, under- and overdosing of general and local anesthetics may be prevented, resulting in favorable hemodynamics and better intra and postoperative pain relieve.

ELIGIBILITY:
Inclusion Criteria:

* any elective surgery under general or neuraxial anesthesia

Exclusion Criteria:

* non elective procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA 1-3 patients presenting for elective surgery under general or neuraxial anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | up to 1 day
  bloodpressure will be compared using conventional techniques and elfitor
Neuraxial block | up to 1 day
  neuraxial block will be compared using conventional techniques and elfitor

SECONDARY OUTCOMES:
Cardiac output | up to 1 day
  during induction of anesthesia the effect of anesthetics or neuraxial blok on cardiac output will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden Medical University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided